CLINICAL TRIAL: NCT03584971
Title: The Effect of Estrogen Levels on Cooperative and Competitive Decision Making and Risk Preferences
Brief Title: Estrogen and Cooperation, Competitiveness, and Risk Preferences
Acronym: FELICIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Frederik Graff, Assistant Professor, RWTH Aachen University
Other Study IDs: 18-053
Record Dates: First submitted 2018-06-21; First posted 2018-07-12 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Behavioral Correlates of Estradiol
Keywords: estradiol; cooperation; competitiveness; risk preferences

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Estradiol via blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- female patients: women in fertility treatment according to Long GnRH Agonist Protocol
- control group: random sample of male students

SUMMARY:
This study observes the effects of female cycle hormones on cooperation, competitiveness and risk preferences under experimental conditions. Especially, the causal effect of estradiol is isolated.

DETAILED DESCRIPTION:
Behavioural theories assume that, as a result of natural selection, women undergo a brief, unconscious change in some psychological aspects during ovulation. This short-term change, "ovulatory shift", is assumed to aim to increase the probability of successful reproduction in the decisive days of the female cycle. Amongst others, it is assumed that women behave particularly uncooperatively and particularly competitively towards other women during the fertile days. Though, empirical evidence is ambiguous.

The effect on risk preferences is unclear. Theory generally assumes that female risk aversion increases in the fertile days. However, empirical studies find partly positive and partly negative correlations.

Within the scope of this study, estradiol levels which are collected in the clinical treatment of patients in the Clinic for Gynaecological Endocrinology and Reproductive Medicine are to be linked with the behavioural economic measures of cooperation, competitiveness, and risk preferences, which are collected using questionnaires or a computer-based decision task.

The aim of the research project is to quasi-experimentally isolate the effect of estradiol on competitiveness, cooperation and risk preferences of women.

No study known to us has ever been able to realize a comparable quasi-experimental design which is necessary to isolate the causal effect of estradiol on different behavioural measures.

In the experimental group, a sample of approx. 50 women in fertility treatment (In Vitro Fertilization/Intracytoplasmic Sperm Injection (IVF/ICSI), long Gonadotropin releasing Hormone (GnRH) agonist protocol) is surveyed. This allows us to create a quasi-experimental design in which the estradiol level is exogenously manipulated and regularly measured.

A random sample of 30 male students of Rheinisch-Westfälische Technische Hochschule (RWTH) Aachen University serves as a control group.

We realize a longitudinal section design with measurement repetitions, which allows inter- and intrapersonal comparisons. A three-stage procedure with two measuring points and a preliminary clarification meeting is planned.

The following measuring instruments are used to record competitiveness, cooperation and risk preference: SOEP Risk Attitude, Social Value Orientation German A, The cooperative and competitive Personality Scale German, Risk aversion, Willingness to compete.

ELIGIBILITY:
Inclusion Criteria:

Patients

1. female
2. patient in fertility treatment according to Long GnRH Agonist Protocol
3. 18 years and older
4. written declaration of consent
5. persons who are contractually capable and mentally able and willing to follow the instructions of the study staff
6. understanding of the German language (written and spoken)

Control group

1. male
2. 18 Years and older
3. written declaration of consent
4. persons who are contractually capable and mentally able and willing to follow the instructions of the study staff
5. understanding of the German language (written and spoken)

Exclusion Criteria:

Patients

1. Illiterate
2. pregnant and breastfeeding women
3. persons who are accommodated in an institution on official or court order
4. persons in a dependent or employment relationship with the auditor
5. simultaneous participation in another clinical trial

Control group

1. Illiterate
2. persons who are accommodated in an institution on official or court order
3. persons in a dependent or employment relationship with the auditor
4. simultaneous participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women in fertility treatment
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of E2 [mg/l] | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of blood concentration of estradiol (E2) in mg/l
Change of LH [mg/l] | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of blood concentration of the luteinizing hormone (LH) in mg/l
Change of Prog [mg/l] | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of blood concentration of progesterone (Prog) in mg/l
Change of Cooperation 1 | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of willingness to cooperate measured via the Social Value Orientation German A (Murphy et al. 2011)
Change of Competitiveness 1 | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of willingness to compete measured via the cooperative and competitive Personality Scale German (Lu et al. 2006)
Change of Risk Preference 1 | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of Risk preferences measured via the SOEP Risk Attitude (DIW Berlin)
Change of Cooperation 2 | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of willingness to cooperate measured via the cooperative and competitive Personality Scale German (Lu et al. 2006)
Change of Competitiveness 2 | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of willingness to compete measured via the Willingness to compete measure based on Niederle & Vesterlund (2007)
Change of Risk Preference 2 | Approx. 10 days after application of GnRH agonist and again approx. 14 days later
  Change of Risk preferences measured via the Risk aversion measure by Holt & Laury (2002)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Rösing, Dr., Principal Investigator — RWTH Aachen
Locations (1):
- RWTH Aachen University Hospital, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranehill, E., Zethraeus, N., Blomberg, L., von Schoultz, B., Hirschberg, A. L., Johannesson, M., & Dreber, A. (2017). Hormonal Contraceptives Do Not Impact Economic Preferences: Evidence from a Randomized Trial. Management Science.
- [Background] Durante, K. M., Griskevicius, V., Hill, S. E., Perilloux, C., & Li, N. P. (2010). Ovulation, female competition, and product choice: Hormonal influences on consumer behavior. Journal of Consumer Research, 37(6), 921-934.
- [Background] Gangestad SW, Thornhill R. Menstrual cycle variation in women's preferences for the scent of symmetrical men. Proc Biol Sci. 1998 May 22;265(1399):927-33. doi: 10.1098/rspb.1998.0380. PMID 9633114
- [Background] Buser, T. (2012a). Digit ratios, the menstrual cycle and social preferences. Games and Economic Behavior, 76(2), 457-470.
- [Background] Buser, T. (2012b). The impact of the menstrual cycle and hormonal contraceptives on competitiveness. Journal of Economic Behavior & Organization, 83(1), 1-10.
- [Background] Wozniak, D., Harbaugh, W. T., & Mayr, U. (2014). The menstrual cycle and performance feedback alter gender differences in competitive choices. Journal of Labor Economics, 32(1), 161-198.
- [Background] Pearson, M., & Schipper, B. C. (2013). Menstrual cycle and competitive bidding. Games and Economic Behavior, 78, 1-20.
- [Background] Drichoutis, A. C., & Nayga, R. M. (2015). Do risk and time preferences have biological roots?. Southern Economic Journal, 82(1), 235-256.
- [Background] Lazzaro SC, Rutledge RB, Burghart DR, Glimcher PW. The Impact of Menstrual Cycle Phase on Economic Choice and Rationality. PLoS One. 2016 Jan 29;11(1):e0144080. doi: 10.1371/journal.pone.0144080. eCollection 2016. PMID 26824245
- [Background] Murphy RO, Ackermann KA. Social value orientation: theoretical and measurement issues in the study of social preferences. Pers Soc Psychol Rev. 2014 Feb;18(1):13-41. doi: 10.1177/1088868313501745. Epub 2013 Sep 23. PMID 24065346
- [Background] Lu S, Au WT, Jiang F, Xie X, Yam P. Cooperativeness and competitiveness as two distinct constructs: validating the Cooperative and Competitive Personality Scale in a social dilemma context. Int J Psychol. 2013;48(6):1135-47. doi: 10.1080/00207594.2012.743666. Epub 2012 Nov 12. PMID 23145818
- [Background] Holt, C. A., & Laury, S. K. (2002). Risk aversion and incentive effects. American economic review, 92(5), 1644-1655.
- [Background] Niederle, M., & Vesterlund, L. (2007). Do women shy away from competition? Do men compete too much?. The Quarterly Journal of Economics, 1067-1101.
- See also: Website of the Deutsches Institut für Wirtschaftsforschung (DIW) Berlin with description and full questionnaires of the German Socio Economic Panel (SOEP) — http://www.diw.de/de/soep